CLINICAL TRIAL: NCT06236230
Title: Basic and Clinical Studies of Levodopa/Carbidopa/Entacapone in the Treatment of Early Parkinson's Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JD-LK2023062-IR01
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; levodopa/carbidopa/entacapone
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa; Stalevo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- levodopa/carbidopa/entacapone (Experimental): levodopa/carbidopa/entacapone is a combination drug consisting of levodopa, carbidopa, and entacapone. Each tablet contains a 1:4 ratio of carbidopa to levodopa and 200 mg of entacapone. The optimum daily dosage of levodopa/carbidopa/entacapone must be determined by careful titration in each patient.
  Interventions: Drug: levodopa/carbidopa/entacapone

INTERVENTIONS:
Drug: levodopa/carbidopa/entacapone — On Day 1, subjects will be treated with levodopa/carbidopa/entacapone. Based on previous regimen. The dosage of levodopa/carbidopa/entacapone will be equal to the previous total daily dose of LD, and the frequency of administration of levodopa/carbidopa/entacapone is three or four times a day.
  Levodopa/carbidopa/entacapone could be titrated in next 2 weeks according to the investigator's judgment, based on individual clinical response and tolerability.
  After 2-week titration, the dose of levodopa/carbidopa/entacapone will remain as constant as possible to the end of study.
  Other Names: Stalevo

SUMMARY:
This is a, open-label, single-arm 8-week investigation of levodopa/carbidopa/entacapone in the treatment of early Parkinson's disease.

DETAILED DESCRIPTION:
This study will enroll subjects who have a diagnosis of PD with Hoehn-Yahr stage 1.5-3.0 and assess the impact of low dosage of levodopa/carbidopa/entacapone treatment on the motor function and quality of life among PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and greater from 30 to 80.
* Diagnosis of idiopathic PD according to the MDS PD Diagnostic Criteria (2015).
* Hoehn-Yahr stage of 1.5-3.0 ("open" stage).
* Not on anti-PD medication or stable on anti-PD medication for at least 30 days.

Exclusion Criteria:

* Diagnosis of atypical Parkinsonian syndrome, vascular Parkinsonism or drug-induced Parkinsonism.
* History of surgery within 6 months.
* Alcoholism, drug abuse, or severe cognitive impairment (including severe Alzheimer's disease)
* Psychiatric illness, epilepsy, pregnancy and breastfeeding, and clinically significant concomitant illnesses
* Participation in another clinical trial within 2 months.
* With dyskinesia.
* Any other condition that, in the opinion of the investigator, makes them ineligible for enrolment.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) III Score | Baseline, Week 8
  The UPDRS is a standardized assessment scale used to measure the patient's disease state. UPDRS Part III measures the motor function of the patient. A higher score indicates greater disability.

SECONDARY OUTCOMES:
Change From Baseline in UPDRS II Score | Baseline, Week 8
  The UPDRS is a standardized assessment scale used to measure the patient's disease state. UPDRS Part II measures the patient's activities of daily living. A higher score indicates greater disability.
Change From Baseline in Health-related Quality of Life Assessed Using the 39-item Parkinson's Disease Questionnaire (PDQ-39) | Baseline, Week 8
  The PDQ-39 instrument is used to assess quality of life in individuals with PD. A lower score indicates better quality of life.
Incidence of dyskinesia and wearing off | Baseline, Week 8
  Dyskinesia and wearing off are common motor complications. A motor complications patient questionnaire will be record.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Feng Liu, MD,PhD, Principal Investigator — Second Affiliated Hospital of Soochow University
Locations (1):
- The Second Affiliated Hospital of Soochow University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Homayoun H. Parkinson Disease. Ann Intern Med. 2018 Sep 4;169(5):ITC33-ITC48. doi: 10.7326/AITC201809040. PMID 30178019
- [Background] Ahlskog JE, Muenter MD. Frequency of levodopa-related dyskinesias and motor fluctuations as estimated from the cumulative literature. Mov Disord. 2001 May;16(3):448-58. doi: 10.1002/mds.1090. PMID 11391738
- [Background] Li J, Lou Z, Liu X, Sun Y, Chen J. Efficacy and Safety of Adjuvant Treatment with Entacapone in Advanced Parkinson's Disease with Motor Fluctuation: A Systematic Meta-Analysis. Eur Neurol. 2017;78(3-4):143-153. doi: 10.1159/000479555. Epub 2017 Aug 16. PMID 28813703
- [Background] Hauser RA, Auinger P; Parkinson Study Group. Determination of minimal clinically important change in early and advanced Parkinson's disease. Mov Disord. 2011 Apr;26(5):813-8. doi: 10.1002/mds.23638. Epub 2011 Mar 24. PMID 21437987
- [Background] Tolosa E, Hernandez B, Linazasoro G, Lopez-Lozano JJ, Mir P, Marey J, Kulisevsky J. Efficacy of levodopa/carbidopa/entacapone versus levodopa/carbidopa in patients with early Parkinson's disease experiencing mild wearing-off: a randomised, double-blind trial. J Neural Transm (Vienna). 2014 Apr;121(4):357-66. doi: 10.1007/s00702-013-1114-x. Epub 2013 Nov 20. PMID 24253234
- [Background] Hauser RA, Panisset M, Abbruzzese G, Mancione L, Dronamraju N, Kakarieka A; FIRST-STEP Study Group. Double-blind trial of levodopa/carbidopa/entacapone versus levodopa/carbidopa in early Parkinson's disease. Mov Disord. 2009 Mar 15;24(4):541-50. doi: 10.1002/mds.22343. PMID 19058133